CLINICAL TRIAL: NCT02781844
Title: An Open-Label, Randomized, Crossover Study to Assess the Pharmacokinetic and Pharmacodynamic Profiles of Once Daily and Twice Daily Dose Regimens of Recombinant Human Parathyroid Hormone (rhPTH[1-84]) Administered Subcutaneously to Subjects With Hypoparathyroidism
Brief Title: Study to Assess the Blood Concentrations and Actions of Recombinant Human Parathyroid Hormone (rhPTH [1-84]) When Given Once and Twice Daily to Participants With Hypoparathyroidism
Acronym: PARALLAX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHP634-101; 2015-004757-40 (EudraCT Number)
Record Dates: First submitted 2016-04-19; First posted 2016-05-25 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A/B or B/A (Experimental): Participants will be randomized to either receive 25 microgram (mcg) rhPTH(1-84) twice daily with no calcium for treatment period 1 and 100mcg rhPTH(1-84) once daily with no calcium for treatment period 2; or 100mcg rhPTH(1-84) once daily with no calcium for treatment period 1 and 25mcg rhPTH(1-84) BID with no calcium for treatment period 2
  Interventions: Drug: 25mcg rhPTH(1-84); Drug: 100mcg rhPTH(1-84)
- C/B or B/C (Experimental): Participants will be randomized to either receive 50mcg rhPTH(1-84) twice daily with no calcium for treatment period 1 and 100mcg rhPTH(1-84) once daily with no calcium for treatment period 2; or 100mcg rhPTH(1-84) once daily with no calcium for treatment period 1 and 50mcg rhPTH(1-84) twice daily with no calcium for treatment period 2
  Interventions: Drug: 50mcg rhPTH(1-84); Drug: 100mcg rhPTH(1-84)
- D/E or E/D (Experimental): Participants will be randomized to either receive 25mcg rhPTH(1-84) twice daily with calcium for treatment period 1 and 100mcg rhPTH(1-84) once daily with calcium for treatment period 2; or 100mcg rhPTH(1-84) once daily with calcium for treatment period 1 and 25mcg rhPTH(1-84) twice daily with calcium for treatment period 2
  Interventions: Drug: 25mcg rhPTH(1-84); Drug: 100mcg rhPTH(1-84)
- F/E or E/F (Experimental): Participants will be randomized to either receive 50mcg rhPTH(1-84) twice daily with calcium for treatment period 1 and 100mcg rhPTH(1-84) once daily with calcium for treatment period 2; or 100mcg rhPTH(1-84) once daily with calcium for treatment period 1 and 50mcg rhPTH(1-84) twice daily with calcium for treatment period 2
  Interventions: Drug: 50mcg rhPTH(1-84); Drug: 100mcg rhPTH(1-84)

INTERVENTIONS:
Drug: 25mcg rhPTH(1-84) — Participants will receive rhPTH(1-84) as twice-daily regimen (12 hours apart) of two 25mcg doses without calcium in cohort 1 and with calcium in cohort 3.
  Other Names: PTH
  Arms: A/B or B/A; D/E or E/D
Drug: 50mcg rhPTH(1-84) — Participants will receive rhPTH(1-84) as twice daily regimen (12 hours apart) of two 50mcg doses without calcium in cohort 2 and with calcium in cohort 4
  Other Names: PTH
  Arms: C/B or B/C; F/E or E/F
Drug: 100mcg rhPTH(1-84) — Participants will receive rhPTH(1-84) as once-daily regimen of one 100 mcg dose without calcium in cohort 1 and 2 and with calcium in cohort 3 and 4 in the morning.
  Other Names: PTH

SUMMARY:
This study is being conducted to characterize the effects of twice daily administration of rhPTH(1-84) on the way the body handles rhPTH(1-84) as well as its actions and safety and tolerability over the course of 24 hours as compared with the current once daily dosing regimen of marketed rhPTH(1-84) (marketed in the United States as Natpara® and in the EU as Natpar).

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
2. Ability to voluntarily provide written, signed, and dated informed consent as applicable to participate in the study.
3. Adult men or women aged greater than or equal (>=) 18 years at the time of consent. The date of participant signature of the informed consent is defined as the beginning of the Screening Period. The Screening Period for this study may encompass both the Administrative Screening Period (if needed) and the Clinical Screening Period. For purposes of this inclusion criterion, age will only be assessed at the time the informed consent is first signed by the study participant.
4. History of hypoparathyroidism for >=12 months, post-diagnosis, inclusive of historical biochemical evidence of hypocalcemia with concomitant serum intact parathyroid hormone (PTH) concentrations below the lower limit of the laboratory normal range.
5. Requirement for supplemental oral calcium treatment >=1000 milligrams (mg) elemental calcium per day.
6. Requirement for therapy with active forms of vitamin D at a minimum dose of >=0.25 microgram (mcg) per day (that is, >=0.25 mcg calcitriol or equivalent per day).
7. Serum calcium level within the laboratory normal reference range based on clinical chemistry lab results at the Clinical Screening Visit (based on central and/or local lab results) and Treatment Period 1, Day -2 (based on central and/or local lab results), or if outside of normal range, considered not clinically significant by the investigator.
8. Urinary calcium excretion >=200mg (5 millimolar [mmol])/24 hour (h), based on a 24-hour collection, collected anytime during the Clinical Screening Period, but prior to check-in to the Clinical Research Center (CRC) at Treatment Period 1, Day -2 (based on central and/or local lab results).
9. Serum magnesium level within the laboratory normal range at the Clinical Screening Visit or, if outside of normal range, considered not clinically significant by the investigator.
10. Serum thyroid function tests within normal laboratory limits at the Clinical Screening Visit, or, if outside of normal range, considered as not clinically significant by the investigator.
11. Serum 25-hydroxyvitamin D (25(OH)D) level between the lower limit of normal and 1.5-fold the laboratory upper limit of normal, or, if outside of this range, considered not clinically significant by the investigator, at the Clinical Screening Visit.
12. Serum creatinine less than (<) 1.5 mg/ decilitre (dL) (<133 micromole [mmol]/ litre [L]) AND estimated creatinine clearance greater than (>) 60 millilitre (mL)/minute (>1.002mL/ Second [s]) at the Clinical Screening Visit, and serum creatinine <1.5 mg/dL (<133mmol/L) at Treatment Period 1, Day -2.
13. Male or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria:

1. Participation in any other investigational drug study in which the last dose of investigational drug occurred within 3 months prior to Day 1 of Treatment Period 1 (or within 5 half-lives, if elimination half-life is greater than 18 days).
2. Presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine (with exception of the condition under study), or neurologic system(s) or psychiatric disease as determined by the investigator.
3. Known history of hypoparathyroidism resulting from an activation mutation in the calcium sensing receptor (CaSR) gene or impaired responsiveness to PTH (pseudohypoparathyroidism).
4. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, including but not limited to, active hyperthyroidism; poorly controlled insulin-dependent diabetes mellitus or type 2 diabetes mellitus; severe and chronic cardiac, liver or renal disease; Cushing's syndrome; neuromuscular disease such as rheumatoid arthritis; myeloma; pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy, bone metastases or a history of skeletal malignancies; primary or secondary hyperparathyroidism; a history of parathyroid carcinoma; hypopituitarism, acromegaly; or multiple endocrine neoplasia types 1 and 2, as determined by the investigator.

5 . In male and female rats, parathyroid hormone caused an increase in the incidence of osteosarcoma (a malignant bone tumor). The occurrence of osteosarcoma was dependent on parathyroid hormone dose and treatment duration. This effect was observed at parathyroid hormone exposure levels ranging from 3 to 71 times the exposure levels in humans receiving a 100 mcg dose of rhPTH(1-84). Therefore, participant who are at increased baseline risk for osteosarcoma such as participant with Paget's disease of bone or unexplained elevations of alkaline phosphatase, pediatric and young adult participants with open epiphyses, participants with hereditary disorders predisposing to osteosarcoma or participant with a prior history of external beam or implant radiation therapy involving the skeleton are excluded.

6. Participants who have a known history of hypercalcemia during initiation of treatment with PTH, PTH analogues or fragments of PTH.

7. Participants who have a known history of hypocalcemia following abrupt withdrawal of treatment with PTH, PTH analogues or fragments of PTH.

8. Participant dependent on regular parenteral calcium infusions (example, calcium gluconate) to maintain calcium homeostasis within 3 months prior to enrollment, as determined by the investigator.

9. Use of the following medications prior to administration of investigational product within: 14 days- thiazide diuretics; 30 days - loop diuretics, lithium, systemic corticosteroids (medical judgment is required by the investigator. Primarily high doses of systemic corticosteroids [example, prednisone] should be excluded. Stable doses of hydrocortisone [example, as treatment for Addison's disease] may be acceptable); 3 months - calcitonin, cinacalcet hydrochloride, treatment with rhPTH(1-84) or N-terminal PTH or PTH-related peptide fragments or analogs; For females: changes in hormone replacement therapy within 3 months are excluded. Stable (>=3 months) hormone replacement therapy is acceptable; 6 months - fluoride tablets, oral bisphosphonates, methotrexate, growth hormone, digoxin, raloxifene or similar selective estrogen receptor modulators (SERMs); 12 months - intravenous bisphosphonates, drug or alcohol abuse, as determined by the investigator.

10. Presence of any clinically significant results from laboratory tests, vital signs assessments, or electrocardiograms (ECGs), as judged by the investigator.

11. Twelve-lead ECG values (average of triplicate readings) demonstrating QTc>450 millisecond (msec) (males) or >470 msec (females) at the Clinical Screening Visit and/or any time points up to and including predose of Day 1 (Period 1).

12. Any medical condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for this study.

13. Positive test result for any of the following viral infections at the Clinical Screening Visit: Hepatitis B surface antigen; hepatitis C; human immunodeficiency virus (HIV) 14. Known significant bleeding diathesis that could preclude multiple venipunctures as determined by the investigator.

15. Participants who have donated a total of 100 mL to 499 mL of whole blood within 30 days prior to dosing, or participants who have donated a total of more than 499 mL of whole blood within 56 days prior to dosing.

16. A positive screen for drugs of abuse at the Clinical Screening Visit, and/or a positive screen for drugs of abuse and alcohol at check-in to the CRC at Treatment Period 1. Participants taking prescription medications that might be detected during the urine screen for drugs of abuse may be enrolled per the investigator's medical judgment.

17. History of a clinically significant illness during the 4 weeks prior to dosing (as determined by the investigator).

18. History of any clinically significant surgery or procedure within the past 8 weeks, as determined by the investigator.

19. History of an allergic response(s) to PTH or PTH analogs, or other clinically significant allergies, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (10):
  - Providence Clinical Research, North Hollywood, California
  - Indiana University, Indianapolis, Indiana
  - University Of Kentucky School of Medicine, Lexington, Kentucky
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - New Orleans Center for Clinical Research (NOCCR) - Knoxville, Knoxville, Tennessee
- CHU de Quebec-Universite Laval, Québec, Canada
- Aarhus Universitetshospital, Aarhus N, Central Jutland, Denmark
- Hungary (3):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Semmelweis Egyetem, Budapest
  - Pécsi Tudományegyetem, Pécs

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in North America and Europe between 04 March 2017 (first participant first visit) to 08 March 2019 (last participant last visit).
Pre-assignment Details: A total of 34 participants were enrolled and 33 completed the study. The study consisted of two treatment periods (Treatment period I and II) with four cohorts. Cohort I included Sequence AB and BA. Cohort II included Sequence CB and BC. Cohort III included Sequence DE and ED, Cohort IV included Sequence FE and EF.
Groups:
- Cohort I: Treatment A / B: Participants received 25 microgram (mcg) rhPTH(1-84) twice daily (BID) with no calcium for treatment period 1 and 100 mcg rhPTH(1-84) once daily (QD) with no calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of greater than or equal to (>=) 5 days but less than or equal to (<=) 30 days between the administration of 25 mcg BID and 100 mcg QD rhPTH(1-84).
- Cohort I: Treatment B / A: Participants received 100 mcg rhPTH(1-84) QD with no calcium for treatment period 1 and 25 mcg rhPTH(1-84) BID with no calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 100 mcg QD and 25 mcg BID rhPTH(1-84).
- Cohort II: Treatment C / B: Participants received 50 mcg rhPTH(1-84) BID with no calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with no calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 50 mcg BID and 100 mcg QD rhPTH(1-84).
- Cohort II: Treatment B / C: Participants received 100 mcg rhPTH(1-84) QD with no calcium for treatment period 1 and 50 mcg rhPTH(1-84) BID with no calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 100 mcg QD and 50 mcg BID rhPTH(1-84).
- Cohort III: Treatment D / E: Participants received 25 mcg rhPTH(1-84) BID with calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 25 mcg BID and 100 mcg QD rhPTH(1-84).
- Cohort III: Treatment E / D: Participants received 100 mcg rhPTH(1-84) QD with calcium for treatment period 1 and 25 mcg rhPTH(1-84) BID with calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 100 mcg QD and 25 mcg BID rhPTH(1-84).
- Cohort IV: Treatment F / E: Participants received 50 mcg rhPTH(1-84) BID with calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 50 mcg BID and 100 mcg QD rhPTH(1-84).
- Cohort IV: Treatment E / F: Participants received 100 mcg rhPTH(1-84) QD with calcium for treatment period 1 and 50 mcg rhPTH(1-84) BID with calcium for treatment period 2 in the morning on Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of 100 mcg QD and 50 mcg BID rhPTH(1-84).
Period: Treatment Period 1
Arm/Group | Cohort I: Treatment A / B | Cohort I: Treatment B / A | Cohort II: Treatment C / B | Cohort II: Treatment B / C | Cohort III: Treatment D / E | Cohort III: Treatment E / D | Cohort IV: Treatment F / E | Cohort IV: Treatment E / F
Started | 5 | 4 | 4 | 4 | 4 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | Cohort I: Treatment A / B | Cohort I: Treatment B / A | Cohort II: Treatment C / B | Cohort II: Treatment B / C | Cohort III: Treatment D / E | Cohort III: Treatment E / D | Cohort IV: Treatment F / E | Cohort IV: Treatment E / F
Started | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included enrolled participants who had received at least 1 dose of rhPTH(1-84).
Groups:
- Cohort I: Treatment A/B or Treatment B/A: Participants received either 25 mcg rhPTH(1-84) BID with no calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with no calcium for treatment period 2; or 100 mcg rhPTH(1-84) QD with no calcium for treatment period 1 and 25 mcg rhPTH(1-84) BID with no calcium for treatment period 2 in the morning of Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of rhPTH(1-84) or the first administration of rhPTH(1-84) in each period for QD or BID dosing, respectively.
- Cohort II: Treatment C/B or Treatment B/C: Participants received either 50 mcg rhPTH(1-84) BID with no calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with no calcium for treatment period 2; or 100 mcg rhPTH(1-84) QD with no calcium for treatment period 1 and 50 mcg rhPTH(1-84) BID with no calcium for treatment period 2 in the morning of Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of rhPTH(1-84) or the first administration of rhPTH(1-84) in each period for QD or BID dosing, respectively.
- Cohort III: Treatment D/E or Treatment E/D: Participants received either 25 mcg rhPTH(1-84) BID with calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with calcium for treatment period 2; or 100 mcg rhPTH(1-84) QD with calcium for treatment period 1 and 25 mcg rhPTH(1-84) BID with calcium for treatment period 2 in the morning of Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of rhPTH(1-84) or the first administration of rhPTH(1-84) in each period for QD or BID dosing, respectively.
- Cohort IV: Treatment F/E or Treatment E/F: Participants receive either 50 mcg rhPTH(1-84) BID with calcium for treatment period 1 and 100 mcg rhPTH(1-84) QD with calcium for treatment period 2; or 100 mcg rhPTH(1-84) QD with calcium for treatment period 1 and 50 mcg rhPTH(1-84) BID with calcium for treatment period 2 in the morning of Day 1 of respective treatment periods. The 2 treatment periods were separated by a washout period of > or = 5 days but < or = 30 days between the administration of rhPTH(1-84) or the first administration of rhPTH(1-84) in each period for QD or BID dosing, respectively.
- Total: Total of all reporting groups
Arm/Group | Cohort I: Treatment A/B or Treatment B/A | Cohort II: Treatment C/B or Treatment B/C | Cohort III: Treatment D/E or Treatment E/D | Cohort IV: Treatment F/E or Treatment E/F | Total
Number analyzed (Participants) | 9 | 8 | 9 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (9.06) | 48.9 (13.48) | 52.4 (13.31) | 45.8 (9.02) | 47.4 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 8 | 7 | 30
  Male | 0 | 2 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 9 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 8 | 8 | 8 | 8 | 32
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time of Maximum Observed Concentration (Cmax) During a Dosing Interval (Tmax) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. Tmax of baseline adjusted rhPTH(1-84) was reported. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Time Frame: QD: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12,16 and 24 hours post-dose ; BID: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12 hours,12 hour 10 minutes,12 hour 20 minutes,12 hour 30 minutes,13 hours, 13 hour 30 minutes,14,16,20,22,24,28 and 36 hours post-dose
Population: Pharmacokinetic (PK) analysis set consisted of all enrolled participants who did not have major protocol violations that affected the validity of the PK results, received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable postdose PK concentration value available for 1 dose regimen.
Measure: Median (Full Range); unit: hours
Groups:
- Cohort I: Treatment A: Participants received 25 mcg rhPTH(1-84) BID with no calcium in the morning on Day 1 of respective treatment period in cohort I.
- Cohort II: Treatment C: Participants received 50 mcg rhPTH(1-84) BID with no calcium in the morning on Day 1 of respective treatment period in Cohort II.
- Cohort I+II: Treatment B: Participants received 100 mcg rhPTH(1-84) QD with no calcium in both cohort I and II in the morning on Day 1 of respective treatment period.
- Cohort III: Treatment D: Participants received 25 mcg rhPTH(1-84) BID with calcium in the morning on Day 1 of respective treatment period in Cohort III.
- Cohort IV: Treatment F: Participants received 50 mcg rhPTH(1-84) BID with calcium in the morning on Day 1 of respective treatment period in Cohort IV.
- Cohort III + IV: Treatment E: Participants received 100 mcg rhPTH(1-84) QD with calcium in both cohort III and IV in the morning on Day 1 of respective treatment period.
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 8 | 15 | 8 | 6 | 14
hours | 7.108 [0.18 to 14.07] | 7.083 [0.17 to 13.50] | 0.333 [0.17 to 4.17] | 1.000 [0.15 to 14.00] | 12.167 [0.17 to 13.50] | 0.667 [0.12 to 4.00]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. Cmax of baseline adjusted rhPTH(1-84) was reported.
Time Frame: QD: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12,16 and 24 hours post-dose; BID: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12 hours,12 hour 10 minutes,12 hour 20 minutes,12 hour 30 minutes,13 hours, 13 hour 30 minutes,14,16,20,22,24,28 and 36 hours post-dose
Population: PK analysis set. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 8 | 15 | 8 | 6 | 14
picogram per milliliter (pg/mL) | 136.9 (50.9) | 213.6 (51.6) | 339.1 (137.8) | 120.9 (83.6) | 100.5 (106.2) | 240.8 (69.6)

3. Primary Outcome: Area Under the Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. AUClast of baseline adjsuted plasma rhPTH(1-84) was reported.
Time Frame: as for outcome 2
Population: PK analysis set. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure and at specific category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram per milliliter (h*pg/mL)
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 8 | 15 | 8 | 6 | 13
hour*picogram per milliliter (h*pg/mL) | 496.0 (34.1) | 653.2 (25.5) | 901.1 (448.5) | 205.0 (106.6) | 261.1 (77.6) | 1044.9 (58.0)

4. Primary Outcome: Area Under the Curve Extrapolated to Infinity (AUCinf) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. AUCinf of baseline adjusted rhPTH(1-84) was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 4 | 7 | 13 | 3 | 1 | 12
h*pg/mL | 484.8 (48.4) | 677.7 (22.9) | 1567.6 (36.7) | 255.0 (198.3) | 600.8 (NA) — Geometric CV% cannot be calculated for one single participant. This outcome measure was analyzed only in one participants for cohort IV. | 1043.5 (50.4)

5. Primary Outcome: Area Under the Concentration Curve From Time Zero to 24 Hours Post the First Dose (AUC0-24) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. AUC0-24 of baseline adjusted rhPTH(1-84) was reported.
Time Frame: QD: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12,16 and 24 hours post-dose; BID: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12 hours,12 hour 10 minutes,12 hour 20 minutes,12 hour 30 minutes,13 hours, 13 hour 30 minutes,14,16,20,22,24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 8 | 15 | 8 | 6 | 13
h*pg/mL | 944.6 (29.9) | 1357.6 (31.3) | 973.7 (334.6) | 577.6 (94.3) | 606.3 (135.3) | 1106.8 (59.3)

6. Primary Outcome: Area Under the Concentration Curve From Time Zero to 12 Hours Post the First Dose (AUC0-12) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. AUC0-12 of baseline adjusted rhPTH(1-84) was reported. AUC(0-12) was planned, analyzed and reported only in participants who received BID treatment ( Treatment A, Treatment C, Treatment D, Treatment F).
Time Frame: BID: Pre-dose,10,20,30 minutes,1,1.5,2,4,8,12 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort III: Treatment D | Cohort IV: Treatment F
Number analyzed (Participants) | 8 | 8 | 8 | 6
h*pg/mL | 462.1 (29.9) | 665.2 (42.3) | 298.8 (113.9) | 220.2 (354.7)

7. Primary Outcome: Area Under the Concentration Curve From Time of the Second Dose to 12 Hours Post the Second Dose (AUC12-24) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. AUC12-24 of baseline adjusted rhPTH(1-84) was reported. AUC(12-24) was planned, analyzed and reported only in participants who received BID treatment ( Treatment A, Treatment C, Treatment D, Treatment F).
Time Frame: BID: 12 hours,12 hour 10 minutes,12 hour 20 minutes,12 hour 30 minutes,13 hours, 13 hour 30 minutes,14,16,20,22,24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort III: Treatment D | Cohort IV: Treatment F
Number analyzed (Participants) | 8 | 8 | 8 | 6
h*pg/mL | 479.0 (33.3) | 679.5 (25.5) | 245.2 (93.5) | 323.2 (71.7)

8. Primary Outcome: Terminal Half-Life (t1/2) of Baseline Adjusted rhPTH(1-84)
Description: Baseline-adjusted rhPTH(1-84) concentrations (participant- and period-specific) were calculated by subtracting baseline endogenous PTH from the raw PTH concentrations. The baseline was defined as premorning-dose endogenous rhPTH(1-84) level on Day 1 for each treatment period. T1/2 of baseline adjusted rhPTH(1-84) was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 4 | 7 | 13 | 3 | 1 | 12
hours | 1.739 (39.461) | 2.073 (38.704) | 1.973 (42.421) | 1.446 (62.293) | 1.773 (NA) — Geometric CV% cannot be calculated for one single participant. This outcome measure was analyzed only in one participant for cohort IV. | 2.190 (38.206)

9. Primary Outcome: Area Under the Concentration-Time Curve That is Above the Baseline, From Time 0 to 24 Hours (AUCabove) of Baseline-Adjusted Serum Calcium Concentrations on Day -1
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. AUCabove of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day -1 was reported. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Time Frame: Day -1
Population: Pharmacodynamic (PD) analysis set consisted of all enrolled participants who did not have major protocol violations that affected the validity of the PD results, received at least 1 dose of rhPTH(1 84) and had at least 1 evaluable post-dose PD value available for 1 dose regimen.
Measure: Mean (Standard Deviation); unit: hour*millimoles per Liter (h*mmol/L)
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 15 | 8 | 6 | 14
hour*millimoles per Liter (h*mmol/L)
  Calcium (Albumin-Corrected) | 2.714 (1.5038) | 1.189 (1.5482) | 0.701 (0.9478) | 0.802 (0.7234) | 1.470 (1.7843) | 0.791 (0.8162)
  Total Calcium | 2.672 (1.8280) | 1.190 (1.3884) | 0.616 (0.8793) | 0.934 (0.7920) | 1.890 (1.7930) | 1.162 (1.2725)

10. Primary Outcome: Area Under the Concentration-Time Curve That is Below the Baseline, From Time 0 to 24 Hours (AUCbelow) of Baseline-Adjusted Serum Calcium Concentrations on Day -1
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. AUCbelow of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day -1 was reported.
Time Frame: Day -1
Population: PD analysis set. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 15 | 8 | 6 | 14
h*mmol/L
  Calcium (Albumin-Corrected) | 0.283 (0.5173) | 0.380 (0.3621) | 1.291 (1.8883) | 0.637 (1.0314) | 0.434 (0.6786) | 0.816 (0.9874)
  Total Calcium | 0.238 (0.4379) | 0.394 (0.3259) | 1.570 (1.9043) | 0.639 (0.9601) | 0.515 (0.6182) | 0.998 (1.3267)

11. Primary Outcome: Time to Maximum Effect (TEmax) of Baseline-Adjusted Serum Calcium Concentrations on Day -1
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. TEmax of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day -1 were reported.
Time Frame: Day -1
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 15 | 8 | 6 | 14
hours
  Calcium (Albumin-Corrected) | 8.000 [4.00 to 16.52] | 13.583 [8.05 to 16.00] | 6.000 [0.00 to 13.80] | 7.317 [3.97 to 23.92] | 9.250 [1.67 to 24.07] | 13.692 [0.00 to 24.73]
  Total Calcium | 8.000 [4.00 to 16.52] | 12.100 [0.00 to 25.47] | 4.200 [0.00 to 16.25] | 5.208 [1.67 to 23.92] | 5.367 [1.67 to 24.07] | 13.692 [0.00 to 24.73]

12. Primary Outcome: Maximum Effect (Emax) of Baseline-Adjusted Serum Calcium Concentrations on Day -1
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. Emax of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day -1 were reported.
Time Frame: Day -1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimoles/Liter (mmol/L)
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 15 | 8 | 6 | 14
millimoles/Liter (mmol/L)
  Calcium (Albumin-Corrected) | 0.284 (0.1495) | 0.110 (0.1098) | 0.102 (0.0892) | 0.098 (0.0539) | 0.148 (0.1398) | 0.107 (0.0783)
  Total Calcium | 0.273 (0.1874) | 0.116 (0.1066) | 0.100 (0.0921) | 0.121 (0.0690) | 0.197 (0.1465) | 0.127 (0.0947)

13. Primary Outcome: Area Under the Concentration-Time Curve That is Above the Baseline, From Time 0 to 24 Hours (AUCabove) of Baseline-Adjusted Serum Calcium Concentrations on Day 1/Day 2
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. AUCabove of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day 1/Day 2 were reported.
Time Frame: Day1- QD: Pre-dose up to 24 hours post dose, Day2- BID: Pre-dose up to 36 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 14
h*mmol/L
  Calcium (albumin-corrected) | 1.222 (1.2757) | 1.084 (0.8887) | 1.645 (1.1038) | 2.860 (4.1108) | 1.468 (1.5533) | 2.610 (1.5520)
  Total Calcium | 1.060 (1.0398) | 0.715 (0.5001) | 1.769 (1.3569) | 3.259 (4.6635) | 1.540 (1.6227) | 2.456 (1.4576)

14. Primary Outcome: Area Under the Concentration-Time Curve That is Below the Baseline, From Time 0 to 24 Hours (AUCbelow) of Baseline-Adjusted Serum Calcium Concentrations on Day 1/Day 2
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. AUCbelow of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day 1/Day 2 was reported.
Time Frame: Day1- QD: Pre-dose up to 24 hours post dose, Day2- BID: Pre-dose up to 36 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 14
h*mmol/L
  Calcium (Albumin-Corrected) | 1.085 (1.1804) | 0.393 (0.6320) | 0.197 (0.2940) | 0.309 (0.5883) | 0.548 (0.6416) | 0.316 (0.5706)
  Total Calcium | 0.944 (1.1352) | 0.362 (0.3115) | 0.320 (0.5456) | 0.273 (0.4174) | 0.601 (0.6863) | 0.437 (0.7870)

15. Primary Outcome: Time to Maximum Effect (TEmax) of Baseline-Adjusted Serum Calcium Concentrations on Day 1/Day 2
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. TEmax of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day 1/Day 2 were reported.
Time Frame: Day1- QD: Pre-dose up to 24 hours post dose, Day2- BID: Pre-dose up to 36 hours post dose
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 14
hours
  Calcium (albumin-corrected) | 11.667 [0.00 to 24.13] | 18.000 [4.00 to 22.00] | 8.017 [1.50 to 24.02] | 18.000 [8.00 to 36.00] | 17.000 [8.10 to 20.00] | 9.075 [0.00 to 16.20]
  Total Calcium | 21.108 [0.00 to 28.02] | 10.000 [1.50 to 22.00] | 9.917 [1.50 to 24.18] | 13.508 [8.00 to 20.00] | 16.000 [8.10 to 36.02] | 8.092 [0.00 to 16.20]

16. Primary Outcome: Maximum Effect (Emax) of Baseline-Adjusted Serum Calcium Concentrations on Day 1/Day 2
Description: Baseline-adjusted concentrations calculated by subtracting the appropriate baseline values from the raw concentrations at each time point. Emax of baseline-adjusted serum calcium (albumin-corrected) and total calcium (calcium [uncorrected]) concentrations on Day 1/Day 2 were reported.
Time Frame: Day1- QD: Pre-dose up to 24 hours post dose, Day2- BID: Pre-dose up to 36 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 14
mmol/L
  Calcium (albumin-corrected) | 0.146 (0.1031) | 0.120 (0.0746) | 0.173 (0.0825) | 0.205 (0.1999) | 0.160 (0.0994) | 0.216 (0.1252)
  Total Calcium | 0.139 (0.1029) | 0.103 (0.0489) | 0.183 (0.0993) | 0.243 (0.2247) | 0.183 (0.0873) | 0.207 (0.1025)

17. Primary Outcome: Total Amount of Urinary Calcium Excretion to Total Relative Amount of Creatinine Over 24 Hours by Day -1
Description: Total amount of urinary calcium excretion to total relative amount of creatinine over 24 hours by Day -1 was reported.
Time Frame: Day -1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol/mmol
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 13
mmol/mmol | 0.806 (0.2284) | 0.836 (0.3020) | 0.727 (0.2859) | 0.874 (0.2670) | 0.855 (0.2858) | 0.807 (0.2764)

18. Primary Outcome: Total Amount of Urinary Calcium Excretion to Total Relative Amount of Creatinine Over 24 Hours by Day 1/ Day 2
Description: Total amount of urinary calcium excretion to total relative amount of creatinine over 24 hours by Day 1/ Day 2 was reported.
Time Frame: Day 1- QD: Pre-dose up to 24 hours post dose, Day 2- BID: Pre-dose up to 24 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimoles Per millimoles (mmol/mmol)
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 14 | 8 | 6 | 14
millimoles Per millimoles (mmol/mmol) | 0.401 (0.1665) | 0.394 (0.1278) | 0.475 (0.1725) | 0.678 (0.2123) | 0.673 (0.2377) | 0.691 (0.2364)

19. Primary Outcome: Total Urinary Excretion of Calcium Over 24 Hours by Day -1
Description: Total urinary excretion of calcium over 24 Hours by Day -1 was reported.
Time Frame: Day -1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 8 | 7 | 15 | 8 | 6 | 13
mmol | 9.348 (3.9559) | 10.239 (3.7130) | 8.880 (3.7407) | 10.831 (2.8306) | 10.735 (2.9224) | 9.717 (2.9354)

20. Primary Outcome: Total Urinary Excretion of Calcium Over 24 Hours by Day 1/ Day 2
Description: Total urinary excretion of calcium over 24 hours by Day1/Day 2 was reported.
Time Frame: Day 1- QD: Pre-dose up to 24 hours post dose, Day 2- BID: Pre-dose up to 24 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 7 | 7 | 14 | 8 | 6 | 14
mmol | 4.904 (1.9684) | 5.137 (1.9800) | 6.037 (2.5353) | 7.440 (2.5379) | 8.813 (2.8213) | 7.928 (2.3159)

21. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE's)
Description: An AE that occured during the study was considered a TEAE if it had a start date/time on or after the first dose of investigational product or if it had a start date before the date of the first dose of investigational product, but increased in severity on or after the date/time of the first dose of investigational product. Number of participants with TEAE's were reported.
Time Frame: From signing of informed consent up to follow up (up to Day 182)
Population: Safety analysis set included enrolled participants who received at least 1 dose of rhPTH(1 84).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
Number analyzed (Participants) | 9 | 8 | 17 | 8 | 8 | 17
Participants | 3 | 1 | 4 | 5 | 3 | 7

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to follow up (up to Day 182)
Description: One participant during the washout out period following the 100 mcg QD dosing treatment period with calcium supplement in cohort III withdrew from the study and considered only in combined arm (Cohort III + IV).
Arm/Group | Cohort I: Treatment A | Cohort II: Treatment C | Cohort I+II: Treatment B | Cohort III: Treatment D | Cohort IV: Treatment F | Cohort III + IV: Treatment E
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/17 | 0/8 | 0/8 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/17 | 0/8 | 0/8 | 0/17
Other Adverse Events (participants affected / at risk) | 3/9 | 1/8 | 4/17 | 5/8 | 3/8 | 7/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I: Treatment A (N=9) | Cohort II: Treatment C (N=8) | Cohort I+II: Treatment B (N=17) | Cohort III: Treatment D (N=8) | Cohort IV: Treatment F (N=8) | Cohort III + IV: Treatment E (N=17)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02781844/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02781844/SAP_001.pdf